CLINICAL TRIAL: NCT06355466
Title: Evaluation of Duration of the Long-term Hemodialysis Catheters Patency and Its Effecting Factors in Chronic Hemodialysis Patients in Golestan Province in 1400-1401
Brief Title: Tunneled Hemodialysis Catheters as Permanent Vascular Access: Evaluating One-year Patency Rate and Affecting Factors
Status: Completed | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Vascular Surgeon, Golestan University of Medical sciences
Other Study IDs: 51-112334
Record Dates: First submitted 2023-12-23; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Vascular Access Devices
Keywords: Hemodialysis; Tunneled catheter; Patency; Antiplatelet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective cross-sectional study, patients with ESRD unfit for AVF/AVG were scheduled for a right or left trans-jugular tunneled catheter placement. All patients were asked about their catheters' function one year after its implantation and the presumed affecting factors on catheters' patency were evaluated.

DETAILED DESCRIPTION:
In this prospective cross-sectional study, the population consisted of patients with end-stage renal failure who were undergoing chronic hemodialysis from 2021-2022 in Golestan province. Patients with end-stage renal failure who were candidates to start or continue dialysis through tunneled catheters as permanent access were included in the study.

According to the 2019 KDOQI guideline, all of the patients were excluded from AVF/ AVG implantation because of one or more of these reasons: heart failure, failed AVF/AVG with no remaining viable option for new AVF/AVG construction, absence of suitable artery/ vein for AVF or AVG construction, patient's preference despite understanding the superiority of AVF/AVG to catheters.

Written informed consent was obtained from all of the patients for conduction and publication of the study.

In all patients, the priority was to insert the catheter through the right jugular unless their right jugular vein was occluded in the preoperative ultrasound, or if it was not possible to pass the wire through the right jugular vein to the right atrium. In these patients, the left jugular vein was used as the insertion site. In some patients left side catheter insertion was not possible as well. These patients whose catheters were placed somewhere else were excluded from the study. In all cases, the proper location of the catheter tip -at the junction of the superior vena cava with the right atrium- was ensured using intraoperative fluoroscopy with a C-arm. For this purpose, catheters of a tip-to-cuff size of 19 and 23 were installed on the right and left side, respectively. For at least one post-implantation session, proper hemodialysis function of the catheter was ensured. All patients underwent surgery by the same vascular surgeon in a single secondary/teaching public center, and due to the restrictions rendered by economic sanctions, a single brand of catheter was used for all patients. A special questionnaire was utilized to record data on age, gender, underlying diseases (diabetes or high blood pressure), medications, and catheter location. All patients' catheter efficacy was re-evaluated one year later by referring to their hemodialysis center or by calling them, and the adequacy of their catheters was recorded to provide adequate flow for hemodialysis. The affecting factors on catheters' patency were evaluated and analysed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

ESRD on chronic hemodialysis Not eligible for AVF/AVG

Exclusion Criteria:

Non-consent of the patient Death Failure to follow up Opportunity for AVF/AVG implantation during the study Failure to implant trans-jugular catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who need continuous hemodialysis and are not eligible to AVF/AVG implantation were scheduled for trans-jugular, tunneled-catheter implantation and after one session of successful hemodialysis were followed one year later for their catheters' function.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
one year patency rate of hemodialysis catheters | one year
  percent of catheters remained patent one year after their implantation

SECONDARY OUTCOMES:
one year patency rate of hemodialysis catheters in age subgroups | one year
  percent of catheters remained patent one year after their implantation in age subgroups
one year patency rate of hemodialysis catheters in diabetic patients | one year
  percent of catheters remained patent one year after their implantation in diabetic patients
one year patency rate of hemodialysis catheters in hypertensive patients | one year
  percent of catheters remained patent one year after their implantation in hypertensive patients
one year patency rate of hemodialysis catheters in patients on antiplatelet drugs | one year
  percent of catheters remained patent one year after their implantation in patients on antiplatelet drugs
one year patency rate of hemodialysis catheters in sex subgroups | one year
  percent of catheters remained patent one year after their implantation in sex subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Pezhman Kharazm, MD, Study Director — assistant professor of vascular surgery
Locations (1):
- Golestan University of Medical Sciences, faculty of medicine, Gorgan, Golestan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thurlow JS, Joshi M, Yan G, Norris KC, Agodoa LY, Yuan CM, Nee R. Global Epidemiology of End-Stage Kidney Disease and Disparities in Kidney Replacement Therapy. Am J Nephrol. 2021;52(2):98-107. doi: 10.1159/000514550. Epub 2021 Mar 22. PMID 33752206
- [Result] Ikizler TA, Cuppari L. The 2020 Updated KDOQI Clinical Practice Guidelines for Nutrition in Chronic Kidney Disease. Blood Purif. 2021;50(4-5):667-671. doi: 10.1159/000513698. Epub 2021 Mar 2. PMID 33652433
- [Result] El Khudari H, Ozen M, Kowalczyk B, Bassuner J, Almehmi A. Hemodialysis Catheters: Update on Types, Outcomes, Designs and Complications. Semin Intervent Radiol. 2022 Feb 18;39(1):90-102. doi: 10.1055/s-0042-1742346. eCollection 2022 Feb. PMID 35210738
- [Result] Boubes K, Shaikh A, Alsauskas Z, Dwyer A. New Directions in Ensuring Catheter Safety. Adv Chronic Kidney Dis. 2020 May;27(3):228-235. doi: 10.1053/j.ackd.2020.02.004. PMID 32891307
- [Result] Obialo CI, Conner AC, Lebon LF. Maintaining patency of tunneled hemodialysis catheters--efficacy of aspirin compared to warfarin. Scand J Urol Nephrol. 2003;37(2):172-6. doi: 10.1080/00365590310008938. PMID 12745728
- [Result] Yaxley J. Haemodialysis catheters - a review of design and function. Expert Rev Med Devices. 2022 Oct;19(10):757-762. doi: 10.1080/17434440.2022.2132148. Epub 2022 Nov 3. PMID 36251438
- [Result] Kumbar L, Yee J. Current Concepts in Hemodialysis Vascular Access Infections. Adv Chronic Kidney Dis. 2019 Jan;26(1):16-22. doi: 10.1053/j.ackd.2018.10.005. PMID 30876612
- [Result] Braet P, Van Holsbeeck A, Buyck PJ, Laenen A, Claes K, De Vusser K, Maleux G. Comparison of Clinical Performance Between Two Types of Symmetric-Tip Hemodialysis Catheters: A Single-Centre, Randomized Trial. Cardiovasc Intervent Radiol. 2023 Aug;46(8):983-990. doi: 10.1007/s00270-023-03476-0. Epub 2023 Jun 13. PMID 37311842
- [Result] Besarab A, Pandey R. Catheter management in hemodialysis patients: delivering adequate flow. Clin J Am Soc Nephrol. 2011 Jan;6(1):227-34. doi: 10.2215/CJN.04840610. Epub 2010 Nov 29. PMID 21115628
- [Result] Agha R, Abdall-Razak A, Crossley E, Dowlut N, Iosifidis C, Mathew G; STROCSS Group. STROCSS 2019 Guideline: Strengthening the reporting of cohort studies in surgery. Int J Surg. 2019 Dec;72:156-165. doi: 10.1016/j.ijsu.2019.11.002. Epub 2019 Nov 6. PMID 31704426
- [Result] Coker MA, Black JR, Li Y, Varma R, Almehmi A, Abdel Aal AK, Gunn AJ. An analysis of potential predictors of tunneled hemodialysis catheter infection or dysfunction. J Vasc Access. 2019 Jul;20(4):380-385. doi: 10.1177/1129729818809669. Epub 2018 Nov 13. PMID 30421638
- [Result] Xiong Y, Yu Y, Yang Y, Wang L, Shi P, Deng Y, Li Y, Fu P. Impacts of age, diabetes, gender, and access type on costs associated with vascular access among Chinese patients on hemodialysis. Int J Artif Organs. 2021 May;44(5):302-309. doi: 10.1177/0391398820962112. Epub 2020 Oct 4. PMID 33016167
- [Result] Valliant AM, Chaudhry MK, Yevzlin AS, Astor B, Chan MR. Tunneled dialysis catheter exchange with fibrin sheath disruption is not associated with increased rate of bacteremia. J Vasc Access. 2015 Jan-Feb;16(1):52-6. doi: 10.5301/jva.5000301. Epub 2014 Sep 2. PMID 25198820
- [Result] Shi M, Cui T, Ma L, Zhou L, Fu P. Catheter Failure and Mortality in Hemodialysis Patients with Tunneled Cuffed Venous Catheters in a Single Center. Blood Purif. 2017;43(4):321-326. doi: 10.1159/000455062. Epub 2017 Jan 31. PMID 28135701
- [Result] Shingarev R, Barker-Finkel J, Allon M. Natural history of tunneled dialysis catheters placed for hemodialysis initiation. J Vasc Interv Radiol. 2013 Sep;24(9):1289-94. doi: 10.1016/j.jvir.2013.05.034. Epub 2013 Jul 18. PMID 23871694
- [Result] Wojtowicz D, Cholewa D, Faba AM, Domanska B, Kokoszka J, Kopacz K, Ficek R, Irzyniec T, Rotkegel SE, Chudek J. Diabetes decreases patency of tunneled catheters in hemodialysis patients after first effective thrombolysis with urokinase. Ren Fail. 2018 Nov;40(1):384-389. doi: 10.1080/0886022X.2018.1487856. PMID 30010473
- [Result] Palmer SC, Di Micco L, Razavian M, Craig JC, Ravani P, Perkovic V, Tognoni G, Graziano G, Jardine M, Pellegrini F, Nicolucci A, Webster A, Strippoli GF. Antiplatelet therapy to prevent hemodialysis vascular access failure: systematic review and meta-analysis. Am J Kidney Dis. 2013 Jan;61(1):112-22. doi: 10.1053/j.ajkd.2012.08.031. Epub 2012 Sep 28. PMID 23022428
- [Result] Yang H, Chen F, Jiao H, Luo H, Yu Y, Hong HG, Li Y, Fu P, Cui T. Management of tunneled-cuffed catheter-related right atrial thrombosis in hemodialysis patients. J Vasc Surg. 2018 Nov;68(5):1491-1498. doi: 10.1016/j.jvs.2018.02.039. Epub 2018 May 24. PMID 29804743
- [Result] Mozafar M, Samsami M, Sobhiyeh MR, Jabbehdari S, Fallah Zavareh M. Effectiveness of aspirin on double lumen permanent catheter efficacy in ESRD. Nephrourol Mon. 2013 Spring;5(2):762-5. doi: 10.5812/numonthly.8733. Epub 2013 Mar 30. PMID 23841041
- [Result] Fry AC, Stratton J, Farrington K, Mahna K, Selvakumar S, Thompson H, Warwicker P. Factors affecting long-term survival of tunnelled haemodialysis catheters--a prospective audit of 812 tunnelled catheters. Nephrol Dial Transplant. 2008 Jan;23(1):275-81. doi: 10.1093/ndt/gfm582. Epub 2007 Sep 21. PMID 17890252
- [Result] Engstrom BI, Horvath JJ, Stewart JK, Sydnor RH, Miller MJ, Smith TP, Kim CY. Tunneled internal jugular hemodialysis catheters: impact of laterality and tip position on catheter dysfunction and infection rates. J Vasc Interv Radiol. 2013 Sep;24(9):1295-302. doi: 10.1016/j.jvir.2013.05.035. Epub 2013 Jul 23. PMID 23891045
- [Result] Weiss MF, Scivittaro V, Anderson JM. Oxidative stress and increased expression of growth factors in lesions of failed hemodialysis access. Am J Kidney Dis. 2001 May;37(5):970-80. doi: 10.1016/s0272-6386(05)80013-7. PMID 11325679